CLINICAL TRIAL: NCT07328802
Title: Clinical Study Protocol for a Single-Center, Prospective, Single-Arm Trial Assessing Icaritin Soft Capsules as Postoperative Adjuvant Therapy in Hepatocellular Carcinoma Patients With High-Risk Factors for Recurrence
Brief Title: Exploration of Sintilimab + Bevacizumab + AG Chemotherapy as First-Line Treatment for Unresectable Advanced/Metastatic Cholangiocarcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHOL-Sintilimab-Bevacizumab-AG
Record Dates: First submitted 2025-06-19; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-06

CONDITIONS: ORR,OS,PFS
MeSH Terms: interventions — Bevacizumab; Albumin-Bound Paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study Cohort (Other)
  Interventions: Drug: Sintilimab combined with bevacizumab and albumin-bound paclitaxel plus gemcitabine

INTERVENTIONS:
Drug: Sintilimab combined with bevacizumab and albumin-bound paclitaxel plus gemcitabine — Patients receive sintilimab (200mg IV Q3W) combined with bevacizumab (15mg/kg IV Q3W) and the AG regimen (albumin-bound paclitaxel + gemcitabine). AG chemotherapy is administered for a total of 8 cycles. After completion of chemotherapy, patients continue sintilimab plus bevacizumab maintenance therapy until disease progression, death, intolerable toxicity, withdrawal of informed consent, initiation of new antitumor therapy, or other protocol-specified reasons for treatment discontinuation, with a maximum treatment duration of 24 months.

SUMMARY:
Evaluation of Efficacy and Safety of Sintilimab Plus Bevacizumab and AG Regimen as First-Line Therapy in Patients with Surgically Ineligible Locally Advanced or Metastatic Cholangiocarcinoma

Objectives:

Primary Objective:

To assess the objective response rate (ORR) as per RECIST v1.1.

Secondary Objectives:

1. To evaluate the disease control rate (DCR) per RECIST v1.1.
2. To determine the duration of response (DOR) per RECIST v1.1.
3. To measure progression-free survival (PFS) per RECIST v1.1.
4. To characterize the safety profile.
5. To determine overall survival (OS) .

Exploratory Objectives:

To investigate potential predictive biomarkers (e.g., PD-L1 expression, tumor mutational burden [TMB]) and their correlation with treatment efficacy (non-mandatory).

DETAILED DESCRIPTION:
This study is a single-arm, Phase II clinical trial evaluating the efficacy and safety of Sintilimab plus Bevacizumab and the AG regimen as first-line therapy in patients with surgically ineligible locally advanced or metastatic cholangiocarcinoma.

After providing informed consent, patients receive:

Sintilimab: 200 mg IV Q3W Bevacizumab: 15 mg/kg IV Q3W AG Chemotherapy: Nab-paclitaxel + Gemcitabine for 8 cycles.

Post-chemotherapy, patients continue Sintilimab + Bevacizumab maintenance until:

Disease progression Death Intolerable toxicity Withdrawal of consent Initiation of new antitumor therapy Other protocol-specified reasons (Maximum treatment duration: 24 months)

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent prior to any trial-related procedures.
2. Male or female aged **≥18 years and ≤75 years**.
3. Histologically or cytologically confirmed, surgically unresectable locally advanced or metastatic cholangiocarcinoma.
4. No prior systemic therapy; subjects who completed postoperative adjuvant therapy **>6 months ago** are eligible.
5. Life expectancy >3 months.
6. At least one measurable lesion per RECIST 1.1 criteria.
7. ECOG PS score 0 or 1.
8. Adequate organ function (all laboratory criteria below must be met):

（1）Absolute neutrophil count (ANC) **≥1.5×10⁹/L** without granulocyte colony-stimulating factor within 14 days; （2）Platelets **≥90×10⁹/L** without transfusion within 14 days; （3）Hemoglobin **>9 g/dL** without transfusion/recombinant erythropoietin within 14 days; （4）Total bilirubin ≤1.5×ULN; （5）AST/ALT ≤2.5×ULN (≤5×ULN allowed if liver metastases present); （6）Serum creatinine ≤1.5×ULN AND creatinine clearance (Cockcroft-Gault formula) **≥60 mL/min**; （7）INR or PT ≤1.5×ULN; （8）TSH within normal range; OR if abnormal, total T3 (or FT3) AND FT4 within normal limits; （9）Cardiac enzymes within normal limits (isolated abnormalities deemed clinically insignificant by investigator are allowed).

9. For women of childbearing potential:

（1）Negative urine/serum pregnancy test within 3 days before Cycle 1 Day 1 (confirm equivocal urine tests with serum testing).

（2）Non-childbearing potential defined as:

1. Postmenopausal (≥1 year amenorrhea), OR
2. Surgically sterilized/hysterectomy. 10. All subjects (regardless of gender) at conception risk must use contraception with <1% annual failure rate during treatment and for 120 days after last dose.

   Exclusion Criteria:
   1. Other malignancies within 5 years prior to first dose (excluding radically cured basal cell carcinoma, squamous cell carcinoma of skin, or carcinoma in situ).
   2. Current participation in interventional clinical trials or receipt of other investigational drugs/devices within 4 weeks before first dose.
   3. Prior therapy with:

   <!-- -->

   1. Anti-PD-1/PD-L1/PD-L2 agents;
   2. Drugs targeting stimulatory/co-inhibitory T-cell receptors (e.g., CTLA-4, OX-40, CD137).

   4. Systemic administration of antitumor Chinese herbal medicines or immunomodulators (e.g., thymosin, interferon, interleukin) within 2 weeks (except localized use for pleural effusion).

   5. Active autoimmune disease requiring systemic treatment within 2 years (e.g., disease-modifying drugs, corticosteroids ≥10 mg/day prednisone equivalent, immunosuppressants).
   1. Exclusions: Hormone replacement (thyroxine/insulin/physiologic steroids);
   2. Known primary immunodeficiency;
   3. Isolated autoantibody positivity requires investigator confirmation of no autoimmune disease.

   6. Systemic glucocorticoids (excluding topical/inhaled) or immunosuppressive therapy within 4 weeks.Note: Physiologic-dose steroids (≤10 mg/day prednisone equivalent) permitted.

   7. Prior anti-angiogenic therapy (e.g., bevacizumab). 8. Active bleeding within 3 months prior to first dose:
   1. Hemoptysis (≥2.5 mL/fresh blood episode);
   2. Gastrointestinal bleeding. 9. High bleeding risk: Tumor invasion of major vessels or radiologist/investigator-assessed bleeding tendency.

   10. Major surgery within 4 weeks (excluding biopsy). 11. Severe unhealed wounds/ulcers/fractures. 12. Aspirin (>325 mg/day) or platelet-inhibiting NSAIDs for >10 consecutive days within 10 days prior to first dose.

   13. Full-dose anticoagulants/thrombolytics for >10 consecutive days within 10 days prior to first dose.Note: Prophylactic low-dose anticoagulants allowed:

   （1）Warfarin ≤1 mg/day (INR ≤1.5); （2）Heparin ≤12,000 U/day; （3）Aspirin ≤100 mg/day. 14. Hereditary bleeding disorders, coagulopathy, or thrombotic history. 15. Clinically uncontrolled pleural effusion/ascites (asymptomatic/minimal fluid without drainage allowed).

   16. Allogeneic organ transplant (excluding corneas) or hematopoietic stem cell transplant.

   17. Hypersensitivity to sintilimab/bevacizumab or excipients. 18. Inadequate recovery from prior intervention toxicities (i.e., >Grade 1 or not returned to baseline, excluding alopecia/fatigue).

   19. HIV infection (HIV 1/2 antibody-positive). 20. Untreated active HBV:
   1. HBsAg-positive AND HBV-DNA > local ULN;
   2. Exceptions:

a. HBV-DNA <500 IU/mL with ongoing antiviral therapy; b. Anti-HBc (+) only with HBV-DNA monitoring. 21. Active HCV infection (HCV antibody-positive AND detectable HCV-RNA). 22. Live attenuated vaccines within 4 weeks prior to first dose. 23. Pregnancy or breastfeeding. 24. Uncontrolled systemic diseases, including:

1. Severe uncontrolled cardiac arrhythmias (e.g., complete LBBB, ≥Grade II AV block, VT/AF);
2. Unstable angina, CHF, NYHA Class ≥II heart failure;
3. Arterial thromboembolism within 6 months (e.g., MI, stroke, TIA);
4. Major surgery/unhealed wounds within 4 weeks; biopsy within 7 days (except IV catheterization);
5. Uncontrolled hypertension (>140/90 mmHg);
6. Active tuberculosis;
7. Uncontrolled systemic infection;
8. Clinical diverticulitis, intra-abdominal abscess, GI obstruction;
9. Decompensated liver disease/active hepatitis;
10. Uncontrolled diabetes (fasting glucose >10 mmol/L);
11. Urine protein ≥++ AND 24-hr urine protein >1.0 g. 25. Psychiatric disorders impairing treatment compliance. 26. Any condition that may:

（1）Interfere with trial results; （2）Prevent full study participation; （3）Pose additional risks (per investigator judgment).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | From baseline (within 28 days prior to enrollment) through disease progression or study completion, up to approximately 2 years.
  Tumor assessments are based on RECIST 1.1. Imaging modalities for this evaluation require:
  Mandatory scans (each cycle):
  Contrast-enhanced CT or MRI of the chest and abdomen
  Baseline assessments (within 28 days ):
  Contrast-enhanced CT/MRI of the pelvis Brain MRI Whole-body bone scan
  Additional baseline imaging if clinically indicated:
  Contrast-enhanced neck CT (if cervical lymphadenopathy present)
  PET/CT protocol:
  Acceptable for baseline screening only Any abnormal findings must undergo confirmatory anatomical imaging (CT/MRI) for target lesion designation

CONTACTS AND LOCATIONS:
Locations (1):
- the Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No